CLINICAL TRIAL: NCT00586430
Title: The Impact of Lorazepam on Cognition in APOE e4 Carriers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Cynthia Stonnington, M.D., Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: 929-05; 929-05
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer's Disease
Keywords: apolipoprotein E e4; Alzheimer's disease; somnolence; Early detection
MeSH Terms: conditions — Alzheimer Disease; Sleepiness | interventions — Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): single 2 mg dose of lorazepam
  Interventions: Drug: lorazepam
- 2 (Placebo Comparator): single dose of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lorazepam — single 2 mg dose of lorazepam
  Other Names: Ativan
  Arms: 1
Drug: placebo — single dose of placebo
  Arms: 2

SUMMARY:
We expect the results of this pilot study to justify a larger study that follows people to determine if certain tests of memory and attention, performed while sleepiness is induced by a single dose of lorazepam (a widely used anti-anxiety medication) could predict an individual's risk of developing AD. We plan to compare cognitively normal people who possess a common gene that increases risk for AD- the apolipoprotein E (APOE) e4 allele-to individuals without this gene. We hypothesize that a single 2 mg dose of lorazepam will cause more cognitive impairment in carriers of the APOE e4 allele than in noncarriers, and that the carriers will recover more slowly from these impairments than noncarriers.

DETAILED DESCRIPTION:
We aim to compare measures of memory and information processing speed at 2.5 hours and 5 hours after the administration of a 2 mg dose of lorazepam or placebo in cognitively normal, 50-65 year old APOE e4 carriers and noncarriers, and determine the differential impact of lorazepam on cognition at each time point. Twenty carriers and 20 noncarriers matched for age, sex, and education will be drawn from a database of persons who have already undergone genotyping for an ongoing study at the Mayo Clinic, excluding people with evidence of depression or cognitive impairment and other medical, neurological or psychiatric conditions. Using a double blind, crossover design, subjects will receive either placebo or a 2 mg dose of lorazepam after baseline testing. Equivalent tests will be repeated 2.5 and 5 hours post challenge. The data analysis will compare APOE e4 carriers to noncarriers.

ELIGIBILITY:
Inclusion Criteria:

* a score of at least 28 on the MMSE
* a score of less than 10 points on the HAM-D-17
* age 50-65
* genotype APOE e3/e4 or APOE e4 non-carriers
* cognitively normal

Exclusion Criteria:

* significant medical, psychiatric, or neurological illnesses
* use of benzodiazepines within the previous four weeks
* currently using sedating antihistamines

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Groton Maze Learning Task | baseline, 2.5 hours and 5 hours

SECONDARY OUTCOMES:
Auditory Verbal Learning Test | baseline, 2.5 hours and 5 hours
1-back test | baseline, 2.5 hours and 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Stonnington, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Stonnington CM, Snyder PJ, Hentz JG, Reiman EM, Caselli RJ. Double-blind crossover study of the cognitive effects of lorazepam in healthy apolipoprotein E (APOE)-epsilon4 carriers. J Clin Psychiatry. 2009 Oct;70(10):1379-84. doi: 10.4088/JCP.08m04593. Epub 2009 Jun 30. PMID 19573495